CLINICAL TRIAL: NCT03405818
Title: An Open-label Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of Kerydin (Registered) (Tavaborole) Topical Solution, 5% In The Treatment Of Onychomycosis Of The Toenail In Pediatric Subjects Ages 6 To 16 Years And 11 Months
Brief Title: An Evaluation of the Safety and Pharmacokinetics of Tavaborole Topical Solution for the Treatment of Fungal Disease of the Toenail in Children and Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAV-ONYC-401; C3371003 (Other: Alias Study Number)
Record Dates: First submitted 2018-01-03; First posted 2018-01-23 (Actual); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Onychomycosis; Tinea Unguium
Keywords: Fungal infection of the nail
MeSH Terms: conditions — Onychomycosis | interventions — tavaborole; Solutions

STUDY DESIGN:
Intervention Model Description: This was a single group study.

ARMS (1):
- Tavaborole 5% Topical Solution (Experimental): All study participants apply study drug
  Interventions: Drug: Tavaborole 5% Topical Solution

INTERVENTIONS:
Drug: Tavaborole 5% Topical Solution — topical solution for application to toenails
  Other Names: Kerydin

SUMMARY:
This was an open-label study to evaluate the safety and pharmacokinetics of tavaborole 5% topical solution in treating distal subungual onychomycosis (a fungal infection) of the toenail in children and adolescents (ages 6 to 16 years).

Following confirmation of eligibility, including laboratory evidence of a fungal organism in the toenail, tavaborole topical solution was applied once daily to all affected toenails for a 48-week treatment period.

Clinical assessment of the extent of infection and safety assessments were performed periodically throughout the 48-week treatment period, and again at 52 weeks (4 weeks after stopping the treatment).

A subgroup of enrolled subjects applied the topical solution to all 10 toenails and a small area of surrounding skin during the first 28 days. These subjects had blood samples analyzed to evaluate the pharmacokinetics (how the drug moves in the body) of tavaborole topical solution in children and adolescents.

DETAILED DESCRIPTION:
This was an open-label study to evaluate the safety, tolerability, and pharmacokinetics of tavaborole 5% topical solution in treating distal subungual onychomycosis (DSO) of the toenail in pediatric subjects aged 6 to 16 years and 11 months. An eligible subject had a target great toenail (TGT) with at least 20% involvement, with a positive potassium hydroxide (KOH) wet mount and positive fungal culture for T. rubrum or T. mentagrophytes.

Eligible subjects applied tavaborole 5% topical solution, once daily to all affected toenails (the TGT as well as all other toenails having the clinical characteristics of onychomycosis) throughout the 48 week treatment period.

Subjects were evaluated at Screening, Baseline (Day 1), and at Weeks 2, 4, 8, 16, 24, 32, 40, 48, and 52. Each evaluation included a clinical assessment of the AEs and local tolerability evaluation.

Additional procedures were performed as follows:

* Mycology sampling at Screening, Week 24, and Week 52/early termination (ET);
* Clinical disease severity of the TGT at Screening, Week 24, and Week 52/ET;
* Safety laboratory testing at Baseline, Week 24, and Week 52/ET;

In this study, there was a PK subgroup of evaluable subjects aged 12 to 16 years and 11 months studied under maximal use conditions. Subjects in this maximal use subgroup applied the study drug on all 10 toenails, including up to 2 mm of the surrounding skin, for 28 days. On Day 15, a predose PK sample was collected to assess steady state trough level. On Day 29, the study drug application was done at the study site, and PK samples were collected prior to dosing, as well as 4, 6, 8, and 24 hours postdose on Days 29 to 30.

ELIGIBILITY:
Inclusion Criteria:

* males or females, ages >/= 6 years and </= 16 years and 11 months
* clinical diagnosis of distal subungual onychomycosis affecting at least 20% of one of the great toenails (target nail); and with positive KOH and positive culture for T. rubrum or T. mentagrophytes from either great toenail

Exclusion Criteria:

* the target toenail has proximal subungual onychomycosis, onychomycosis involving the nail lunula, superficial white onychomycosis, dermatophytoma, exclusively lateral disease, or yellow or brown spikes, or has co-infection with certain fungi or molds
* anatomic abnormalities of the toes or toenail
* current or past history of chronic moccasin-type tinea pedis
* current or past history of psoriasis or lichen planus
* history of significant chronic fungal disease (other than onychomycosis)
* diabetes
* immunodeficiency

Ages: 72 Months to 203 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Madera Family Medical Group, Madera, California
  - Stanford University School of Medicine, Palo Alto, California
  - MedStar Health Research Institute - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Doctors Research Network, South Miami, Florida
  - University Hospital, SUNY Downstate Medical Center, Brooklyn, New York
  - Skin Specialty Dermatology, New York, New York
  - Cyn3rgy Research, Gresham, Oregon
  - Oregon Dermatology & Research Center, Portland, Oregon
  - West Houston Clinical Research Services LLC, Houston, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Jordan Valley Dermatology Center, West Jordan, Utah
  - PI Coor Clinical Research, LLC, Burke, Virginia

REFERENCES:
- [Derived] Rich P, Spellman M, Purohit V, Zang C, Crook TJ. Tavaborole 5% Topical Solution for the Treatment of Toenail Onychomycosis in Pediatric Patients: Results from a Phase 4 Open-Label Study. J Drugs Dermatol. 2019 Feb 1;18(2):190-195. PMID 30811142

RESULTS

PARTICIPANT FLOW:
Groups:
- Kerydin: Participants applied Kerydin (tavaborole) 5 percent solution, topically once daily for 48 weeks and followed up to 4 weeks after last dose of study drug.
Period: Overall Study
Arm/Group | Kerydin
Started | 55
Completed | 47
Not Completed | 8
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 confirmed dose of study drug and had at least 1 post-baseline safety assessment.
Arm/Group | Kerydin
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.2 (2.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local Tolerability Reactions by Severity
Description: Local tolerability reactions consisted of burning/stinging, induration/edema, oozing and crusting, pruritus, erythema, and scaling. Here 0 indicates None, 1 (Mild), 2 (Moderate) and 3 (severe). Grading details are as follows: Burning/Stinging (0: no stinging/burning, 1: slight warm, 2: definite warm, 3: hot); Induration/Edema (0: no elevation, 1: barely perceptible elevation, 2: clearly perceptible elevation but not extensive, 3: marked and extensive elevation); Oozing and Crusting (0: absent, 1: faint signs of oozing, 2: definite oozing, 3: marked and extensive oozing); Pruritus (0: no pruritus, 1: occasional, slight itching, 2: constant itching which is not disturbing sleep, 3: severe bothersome itching/scratching which is disturbing sleep); Erythema (0: no redness present, 1: faintly detectable erythema; very light pink, 2: dull red, 3: deep/dark red); Scaling (0: no scaling, 1: barely perceptible shedding, 2: obvious but not profuse scaling, 3: heavy scale production).
Time Frame: Baseline up to Week 52
Population: Safety Population: all participants who received at least 1 confirmed dose of study drug and had at least 1 post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Kerydin
Number analyzed (Participants) | 54
Participants
  None Burning/Stinging | 54
  Mild Burning/Stinging | 0
  Moderate Burning/Stinging | 1
  Severe Burning/Stinging | 0
  None Induration/Edema | 53
  Mild Induration/Edema | 4
  Moderate Induration/Edema | 2
  Severe Induration/Edema | 1
  None Oozing and Crusting | 54
  Mild Oozing and Crusting | 2
  Moderate Oozing and Crusting | 1
  Severe Oozing and Crusting | 0
  None Pruritus | 53
  Mild Pruritus | 2
  Moderate Pruritus | 1
  Severe Pruritus | 0
  None Erythema | 50
  Mild Erythema | 6
  Moderate Erythema | 2
  Severe Erythema | 0
  None Scaling | 51
  Mild Scaling | 4
  Moderate Scaling | 3
  Severe Scaling | 1

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both serious and non-serious AEs.
Time Frame: Baseline up to 28 days after last dose of study drug (up to Week 52)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Kerydin
Number analyzed (Participants) | 54
Participants
  Participants with AEs | 30
  Participants with SAEs | 1

3. Primary Outcome: Number of Participants With Adverse Events (AEs) By Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs were classified as mild, moderate and severe based on severity assessment by investigator and defined as: Mild = symptoms barely noticeable to the participant or does not make the participant uncomfortable; moderate = symptoms of a sufficient severity to make the participant uncomfortable; severe = symptoms of a sufficient severity to cause the participant severe discomfort.
Time Frame: Baseline up to 28 days after last dose of study drug (up to Week 52)
Population: Safety Population: all participants who received at least 1 confirmed dose of study drug and had at least 1 post-baseline safety assessment. Here, "N" signifies number of participants evaluable for this specified outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Kerydin
Number analyzed (Participants) | 30
Participants
  Mild | 12
  Moderate | 16
  Severe | 2

4. Primary Outcome: Change From Baseline in Hematology Parameters (Leukocytes: Basophils, Eosinophils, Lymphocytes, Monocytes and Neutrophils) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of leukocytes
Arm/Group | Kerydin
Number analyzed (Participants) | 54
percentage of leukocytes
  Baseline: Basophils/Leukocytes: number analyzed (Participants) | 49
  Baseline: Basophils/Leukocytes | 0.6 (0.53)
  Baseline: Eosinophil/Leukocytes: number analyzed (Participants) | 49
  Baseline: Eosinophil/Leukocytes | 3.3 (2.30)
  Baseline: Lymphocytes/Leukocytes: number analyzed (Participants) | 49
  Baseline: Lymphocytes/Leukocytes | 34.4 (8.89)
  Baseline: Monocytes/Leukocytes: number analyzed (Participants) | 49
  Baseline: Monocytes/Leukocytes | 6.8 (2.12)
  Baseline: Neutrophils/Leukocytes: number analyzed (Participants) | 49
  Baseline: Neutrophils/Leukocytes | 55.1 (9.77)
  Change at Week 24: Basophils/Leukocytes: number analyzed (Participants) | 42
  Change at Week 24: Basophils/Leukocytes | 0.1 (0.67)
  Change at Week 24: Eosinophil/Leukocytes: number analyzed (Participants) | 42
  Change at Week 24: Eosinophil/Leukocytes | -0.5 (2.31)
  Change at Week 24: Lymphocytes/Leukocytes: number analyzed (Participants) | 42
  Change at Week 24: Lymphocytes/Leukocytes | 1.1 (9.34)
  Change at Week 24: Monocytes/Leukocytes: number analyzed (Participants) | 42
  Change at Week 24: Monocytes/Leukocytes | -0.2 (2.00)
  Change at Week 24: Neutrophils/Leukocytes: number analyzed (Participants) | 42
  Change at Week 24: Neutrophils/Leukocytes | -0.7 (10.33)

5. Primary Outcome: Change From Baseline in Hematology Parameters (Leukocytes: Basophils, Eosinophils, Lymphocytes, Monocytes and Neutrophils) at Week 52
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of leukocytes
Arm/Group | Kerydin
Number analyzed (Participants) | 43
percentage of leukocytes
  Change at Week 52: Basophils/Leukocytes | 0.1 (0.60)
  Change at Week 52: Eosinophils/Leukocytes | 0.3 (2.82)
  Change at Week 52: Lymphocytes/Leukocytes | 0.7 (7.91)
  Change at Week 52: Monocytes/Leukocytes | -0.5 (1.93)
  Change at Week 52: Neutrophils/Leukocytes | -0.7 (9.64)

6. Primary Outcome: Change From Baseline in Hematology Parameter (Hematocrit) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: volume percentage of red blood cells
Arm/Group | Kerydin
Number analyzed (Participants) | 54
volume percentage of red blood cells
  Baseline: number analyzed (Participants) | 49
  Baseline | 42.04 (3.460)
  Change at Week 24: number analyzed (Participants) | 42
  Change at Week 24 | 0.57 (2.534)

7. Primary Outcome: Change From Baseline in Hematology Parameter (Hematocrit) at Week 52
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: volume percentage of red blood cells
Arm/Group | Kerydin
Number analyzed (Participants) | 43
volume percentage of red blood cells | -0.12 (1.838)

8. Primary Outcome: Change From Baseline in Hematology Parameter (Erythrocytes) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Kerydin
Number analyzed (Participants) | 54
10^12 cells per liter
  Baseline: number analyzed (Participants) | 49
  Baseline | 4.786 (0.4323)
  Change at Week 24: number analyzed (Participants) | 42
  Change at Week 24 | 0.045 (0.2522)

9. Primary Outcome: Change From Baseline in Hematology Parameter (Erythrocytes) at Week 52
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Kerydin
Number analyzed (Participants) | 43
10^12 cells per liter | -0.009 (0.2004)

10. Primary Outcome: Change From Baseline in Hematology Parameters (Hemoglobin) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gram per deciliter (g/dL)
Arm/Group | Kerydin
Number analyzed (Participants) | 54
gram per deciliter (g/dL)
  Baseline: number analyzed (Participants) | 49
  Baseline | 13.79 (1.138)
  Change at Week 24: number analyzed (Participants) | 42
  Change at Week 24 | 0.11 (0.650)

11. Primary Outcome: Change From Baseline in Hematology Parameters (Hemoglobin) at Week 52
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: gram per deciliter (g/dL)
Arm/Group | Kerydin
Number analyzed (Participants) | 43
gram per deciliter (g/dL) | 0.06 (0.637)

12. Primary Outcome: Change From Baseline in Hematology Parameters (Leukocytes and Platelets) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Kerydin
Number analyzed (Participants) | 54
10^9 cells per liter
  Baseline: Leukocytes: number analyzed (Participants) | 49
  Baseline: Leukocytes | 7.11 (1.723)
  Baseline: Platelets: number analyzed (Participants) | 49
  Baseline: Platelets | 255.6 (49.90)
  Change at Week 24: Leukocytes: number analyzed (Participants) | 42
  Change at Week 24: Leukocytes | -0.51 (1.716)
  Change at Week 24: Platelets: number analyzed (Participants) | 42
  Change at Week 24: Platelets | -4.1 (32.62)

13. Primary Outcome: Change From Baseline in Hematology Parameters (Leukocytes and Platelets) at Week 52
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Kerydin
Number analyzed (Participants) | 43
10^9 cells per liter
  Change at Week 52: Leukocytes | -0.62 (1.940)
  Change at Week 52: Platelets | -9.4 (31.23)

14. Primary Outcome: Change From Baseline in Chemistry Parameters (Alanine Aminotransferase, Alkaline Phosphatase and Aspartate Aminotransferase) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: International Unit per liter (IU/L)
Arm/Group | Kerydin
Number analyzed (Participants) | 54
International Unit per liter (IU/L)
  Baseline: Alanine Aminotransferase | 14.6 (8.23)
  Baseline: Alkaline Phosphatase | 178.7 (90.33)
  Baseline: Aspartate Aminotransferase | 21.7 (17.60)
  Change at Week 24:Alanine Aminotransferase: number analyzed (Participants) | 50
  Change at Week 24:Alanine Aminotransferase | -1.7 (8.21)
  Change at Week 24:Alkaline Phosphatase: number analyzed (Participants) | 50
  Change at Week 24:Alkaline Phosphatase | -1.5 (42.81)
  Change at Week 24:Aspartate Aminotransferase: number analyzed (Participants) | 50
  Change at Week 24:Aspartate Aminotransferase | -3.3 (17.52)

15. Primary Outcome: Change From Baseline in Chemistry Parameters (Alanine Aminotransferase, Alkaline Phosphatase and Aspartate Aminotransferase) at Week 52
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: International Unit per liter (IU/L)
Arm/Group | Kerydin
Number analyzed (Participants) | 47
International Unit per liter (IU/L)
  Change at Week 52:Alanine Aminotransferase | -1.6 (11.32)
  Change at Week 52:Alkaline Phosphatase | -18.4 (60.10)
  Change at Week 52:Aspartate Aminotransferase | -2.7 (19.87)

16. Primary Outcome: Change From Baseline in Chemistry Parameters (Albumin and Protein) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gram per deciliter (g/dL)
Arm/Group | Kerydin
Number analyzed (Participants) | 54
gram per deciliter (g/dL)
  Baseline: Albumin | 4.49 (0.250)
  Baseline: Protein | 6.94 (0.395)
  Change at Week 24: Albumin: number analyzed (Participants) | 50
  Change at Week 24: Albumin | -0.05 (0.374)
  Change at Week 24: Protein: number analyzed (Participants) | 50
  Change at Week 24: Protein | -0.04 (0.502)

17. Primary Outcome: Change From Baseline in Chemistry Parameters (Albumin and Protein) at Week 52
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: gram per deciliter (g/dL)
Arm/Group | Kerydin
Number analyzed (Participants) | 47
gram per deciliter (g/dL)
  Change at Week 52: Albumin | -0.08 (0.375)
  Change at Week 52: Protein | -0.07 (0.492)

18. Primary Outcome: Change From Baseline in Chemistry Parameters (Bilirubin, Creatinine, Glucose [Non-fasting] and Urea Nitrogen) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Kerydin
Number analyzed (Participants) | 54
milligram per deciliter (mg/dL)
  Baseline: Bilirubin | 0.46 (0.279)
  Baseline: Creatinine | 0.68 (0.150)
  Baseline: Glucose [non-fasting] | 87.5 (11.65)
  Baseline: Urea Nitrogen | 13.5 (3.12)
  Change at Week 24: Bilirubin: number analyzed (Participants) | 50
  Change at Week 24: Bilirubin | 0.03 (0.141)
  Change at Week 24: Creatinine: number analyzed (Participants) | 50
  Change at Week 24: Creatinine | 0.01 (0.122)
  Change at Week 24: Glucose [non-fasting]: number analyzed (Participants) | 50
  Change at Week 24: Glucose [non-fasting] | 0.0 (15.15)
  Change at Week 24: Urea Nitrogen: number analyzed (Participants) | 50
  Change at Week 24: Urea Nitrogen | -0.1 (3.55)

19. Primary Outcome: Change From Baseline in Chemistry Parameters (Bilirubin, Creatinine, Glucose [Non-fasting] and Urea Nitrogen) at Week 52
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Kerydin
Number analyzed (Participants) | 47
milligram per deciliter (mg/dL)
  Change at Week 52: Bilirubin | -0.01 (0.155)
  Change at Week 52: Creatinine | 0.04 (0.124)
  Change at Week 52: Glucose [non-fasting] | 5.9 (19.61)
  Change at Week 52: Urea Nitrogen | -0.7 (2.93)

20. Primary Outcome: Change From Baseline in Chemistry Parameters (Potassium and Sodium) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Kerydin
Number analyzed (Participants) | 54
millimole per liter (mmol/L)
  Baseline: Potassium | 4.25 (0.404)
  Baseline: Sodium | 138.0 (1.95)
  Change at Week 24: Potassium: number analyzed (Participants) | 50
  Change at Week 24: Potassium | -0.05 (0.444)
  Change at Week 24: Sodium: number analyzed (Participants) | 50
  Change at Week 24: Sodium | 1.6 (2.29)

21. Primary Outcome: Change From Baseline in Chemistry Parameters (Potassium and Sodium) at Week 52
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Kerydin
Number analyzed (Participants) | 47
millimole per liter (mmol/L)
  Change at Week 52: Potassium | 0.00 (0.473)
  Change at Week 52: Sodium | 2.1 (2.83)

22. Primary Outcome: Change From Baseline in Vital Sign (Blood Pressure) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Kerydin
Number analyzed (Participants) | 54
millimeter of mercury (mmHg)
  Baseline: Systolic Blood Pressure | 110.9 (11.65)
  Baseline: Diastolic Blood Pressure | 68.3 (7.92)
  Change at Week 24: Systolic Blood Pressure: number analyzed (Participants) | 50
  Change at Week 24: Systolic Blood Pressure | 0.4 (10.02)
  Change at Week 24: Diastolic Blood Pressure: number analyzed (Participants) | 50
  Change at Week 24: Diastolic Blood Pressure | 1.0 (9.34)

23. Primary Outcome: Change From Baseline in Vital Sign (Blood Pressure) at Week 52
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Kerydin
Number analyzed (Participants) | 47
millimeter of mercury (mmHg)
  Change at Week 52: Systolic Blood Pressure | 0.1 (9.52)
  Change at Week 52: Diastolic Blood Pressure | 1.0 (7.61)

24. Primary Outcome: Change From Baseline in Vital Sign (Pulse Rate) at Week 24
Description: Pulse rate was defined as the number of pulsations noted in a peripheral artery per minute after participant rested supine for 5 minutes.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Kerydin
Number analyzed (Participants) | 54
Beats per minute (bpm)
  Baseline | 76.2 (14.39)
  Change at Week 24: number analyzed (Participants) | 50
  Change at Week 24 | -3.0 (10.49)

25. Primary Outcome: Change From Baseline in Vital Sign (Pulse Rate) at Week 52
Description: as for outcome 24
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Kerydin
Number analyzed (Participants) | 47
Beats per minute (bpm) | -3.9 (10.66)

26. Primary Outcome: Change From Baseline in Vital Sign (Respiratory Rate) at Week 24
Description: Respiratory rate was defined as the number of inspirations per minute.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Kerydin
Number analyzed (Participants) | 54
Breaths per minute
  Baseline | 16.1 (2.37)
  Change at Week 24: number analyzed (Participants) | 50
  Change at Week 24 | 0.2 (2.62)

27. Primary Outcome: Change From Baseline in Vital Sign (Respiratory Rate) at Week 52
Description: Respiratory rate was defined as the number of inspirations per minute.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Kerydin
Number analyzed (Participants) | 47
Breaths per minute | -0.5 (2.77)

28. Primary Outcome: Percentage of Participants With Complete Cure of Target Great Toenail (TGT) at Week 52
Description: Complete cure was defined as completely clear nail, negative fungal culture and negative potassium hydroxide (KOH) wet mount.
Time Frame: Week 52
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Kerydin
Number analyzed (Participants) | 47
percentage of participants | 8.5

29. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Tavaborole
Time Frame: Pre-dose, 4, 6, 8, 24 hours post-dose on Day 29
Population: Pharmacokinetics (PK) population: all participants from the maximal use subgroup (aged between 12 to 16 years and 11 months with once daily application to all 10 toenails, including up to 2 millimeter [mm] of the surrounding skin) and had PK data available.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Kerydin
Number analyzed (Participants) | 37
Nanogram per milliliter (ng/mL) | 5.4049 (4.32509)

30. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Tavaborole
Time Frame: Pre-dose, 4, 6, 8, 24 hours post-dose on Day 29
Population: Pharmacokinetics (PK) population: all participants from the maximal use subgroup (aged between 12 to 16 years and 11 months with once daily application to all 10 toenails, including up to 2 millimeter [mm] of the surrounding skin) and had PK data available. Here, "N" signifies number of participants evaluable for this specified outcome measure.
Measure: Median (Full Range); unit: hour
Arm/Group | Kerydin
Number analyzed (Participants) | 36
hour | 6.000 [0.00 to 24.20]

31. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Hour Zero to Hour 24 (AUC24) of Tavaborole
Description: AUC24 was defined as the area under the plasma concentration-time curve from hour 0 to hour 24. AUC24 was calculated using the linear trapezoidal rule.
Time Frame: Pre-dose, 4, 6, 8, 24 hours post-dose on Day 29
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Kerydin
Number analyzed (Participants) | 15
hour*nanogram per milliliter (hr*ng/mL) | 102.273 (60.9282)

32. Secondary Outcome: Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUCinf) of Tavaborole
Time Frame: Pre-dose, 4, 6, 8, 24 hours post-dose on Day 29
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Kerydin
Number analyzed (Participants) | 15
hour*nanogram per milliliter (hr*ng/mL) | 124.820 (73.5924)

33. Secondary Outcome: Elimination Rate Constant of Tavaborole
Description: Elimination rate constant was defined as the rate at which a drug was removed from the body.
Time Frame: Pre-dose, 4, 6, 8, 24 hours post-dose on Day 29
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: per hour
Arm/Group | Kerydin
Number analyzed (Participants) | 15
per hour | 0.08528 (0.024508)

34. Secondary Outcome: Elimination Half-Life of Tavaborole
Description: Elimination half-life (t1/2) was defined as the time required for the body to eliminate half of the drug than its original concentration.
Time Frame: Pre-dose, 4, 6, 8, 24 hours post-dose on Day 29
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Kerydin
Number analyzed (Participants) | 15
hour | 9.783 (7.1245)

35. Secondary Outcome: Percentage of Participants With Almost Complete Cure of Target Great Toenail (TGT) at Week 24 and 52
Description: Almost complete cure was defined as almost clear nail and negative mycology (negative mycology was defined as negative fungal culture and negative KOH wet mount).
Time Frame: Week 24, 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Kerydin
Number analyzed (Participants) | 54
percentage of participants
  Week 24: number analyzed (Participants) | 50
  Week 24 | 10
  Week 52: number analyzed (Participants) | 47
  Week 52 | 14.9

36. Secondary Outcome: Percentage of Participants With Clinical Efficacy of Target Great Toenail (TGT) at Week 24 and 52
Description: Clinical efficacy target great toenail (TGT) was defined as completely clear nail or almost clear nail.
Time Frame: Week 24, 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Kerydin
Number analyzed (Participants) | 54
percentage of participants
  Week 24: number analyzed (Participants) | 50
  Week 24 | 10
  Week 52: number analyzed (Participants) | 47
  Week 52 | 25.5

37. Secondary Outcome: Percentage of Participants With Mycological Cure of Target Great Toenail (TGT) at Week 24 and 52
Description: Mycological cure was defined as negative mycology of the TGT. Negative mycology was defined as negative fungal culture and negative potassium hydroxide (KOH) wet mount. Participants with only one result for either fungal culture or KOH were excluded from this analysis.
Time Frame: Week 24, 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Kerydin
Number analyzed (Participants) | 54
percentage of participants
  Week 24: number analyzed (Participants) | 50
  Week 24 | 38.0
  Week 52: number analyzed (Participants) | 47
  Week 52 | 36.2

38. Secondary Outcome: Percentage of Participants With Negative Fungal Culture of the Target Great Toenail (TGT) at Weeks 24 and 52
Time Frame: Week 24, 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Kerydin
Number analyzed (Participants) | 54
percentage of participants
  Week 24: number analyzed (Participants) | 50
  Week 24 | 96
  Week 52: number analyzed (Participants) | 47
  Week 52 | 87.2

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Adverse events were collected for safety population.
Arm/Group | Kerydin
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 1/54
Other Adverse Events (participants affected / at risk) | 30/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Kerydin (N=54)
Appendicitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Kerydin (N=54)
Nasopharyngitis (Infections and infestations) | 7
Sinusitis (Infections and infestations) | 3
Influenza (Infections and infestations) | 2
Acute sinusitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Hand-foot-and-mouth disease (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 5
Concussion (Injury, poisoning and procedural complications) | 2
Arthropod sting (Injury, poisoning and procedural complications) | 1
Eye injury (Injury, poisoning and procedural complications) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Aphthous stomatitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Headache (Nervous system disorders) | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Application site erythema (General disorders) | 1
Blood iron decreased (Investigations) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT03405818/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT03405818/SAP_001.pdf